CLINICAL TRIAL: NCT00002529
Title: Adjuvant Therapy for Post/Perimenopausal Patients With Node Positive Breast Cancer Who Are Suitable for Endocrine Therapy Alone.
Brief Title: Hormone Therapy and Chemotherapy in Treating Perimenopausal or Postmenopausal Women With Node-Positive Breast Cancer
Acronym: 12-93
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ETOP IBCSG Partners Foundation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000078385; IBCSG-12-93 (Other: International Breast Cancer Study Group); EU-93015; NCI-F93-0010
Record Dates: First submitted 1999-11-01; First posted 2004-07-29 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2012-07

CONDITIONS: Breast Cancer
Keywords: stage II breast cancer; stage IIIA breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Cyclophosphamide; Doxorubicin; Epirubicin; Tamoxifen; Toremifene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- AC with concurrent tamoxifen (Experimental): AC for 4 cycles with concurrent tamoxifen for 5 years
  Interventions: Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: epirubicin hydrochloride; Drug: tamoxifen citrate
- AC followed by tamoxifen (Experimental): AC for 4 cycles followed by tamoxifen to 5 years from randomization.
  Interventions: Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: epirubicin hydrochloride; Drug: tamoxifen citrate
- Tamoxifen alone (Experimental): Tamoxifen alone for 5 years.
  Interventions: Drug: tamoxifen citrate
- AC with concurrent toremifene (Experimental): AC for 4 cycles with concurrent toremifene for 5 years.
  Interventions: Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: epirubicin hydrochloride; Drug: toremifene
- AC followed by toremifene (Experimental): AC for 4 cycles followed by toremifene to 5 years from randomization.
  Interventions: Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: epirubicin hydrochloride; Drug: toremifene
- Toremifene alone (Experimental): Toremifene alone for 5 years.
  Interventions: Drug: toremifene

INTERVENTIONS:
Drug: cyclophosphamide — cyclophosphamide 600 mg/m2 i.v. day 1) every 21 days
  Arms: AC followed by tamoxifen; AC followed by toremifene; AC with concurrent tamoxifen; AC with concurrent toremifene
Drug: doxorubicin hydrochloride — doxorubicin 60 mg/m2 i.v. day 1) every 21 days, intravenous.
  Arms: AC followed by tamoxifen; AC followed by toremifene; AC with concurrent tamoxifen; AC with concurrent toremifene
Drug: epirubicin hydrochloride — epirubicin 90 mg/m2 i.v. day 1) every 21 days, intravenous.
  Arms: AC followed by tamoxifen; AC followed by toremifene; AC with concurrent tamoxifen; AC with concurrent toremifene
Drug: tamoxifen citrate — Tamoxifen 20 mg daily.
  Arms: AC followed by tamoxifen; AC with concurrent tamoxifen; Tamoxifen alone
Drug: toremifene — Toremifene 60 mg daily.
  Arms: AC followed by toremifene; AC with concurrent toremifene; Toremifene alone

SUMMARY:
RATIONALE: Estrogen can stimulate the growth of breast cancer cells. Hormone therapy may fight breast cancer by blocking the uptake of estrogen. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy with hormone therapy may kill more tumor cells. It is not yet known which treatment regimen is more effective for breast cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of hormone therapy during or after combination chemotherapy or hormone therapy alone in treating perimenopausal or postmenopausal women who have stage II or stage IIIA breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare overall survival and local and systemic disease-free survival produced by adjuvant chemoendocrine therapy with 4 courses of anthracycline/cyclophosphamide and concurrent vs. sequential tamoxifen (TMX) or toremifene (TOR) in peri- and postmenopausal women with node-positive breast cancer who are considered suitable for endocrine therapy alone. II. Evaluate these same endpoints in patients randomized to chemoendocrine therapy vs. endocrine therapy alone. III. Evaluate these same endpoints in patients randomized to TMX vs. TOR as the endocrine therapy agent. IV. Compare the quality of life of patients treated on these regimens. V. Compare the toxic effects of these regimens.

OUTLINE: This is a randomized study. Patients are stratified by type of primary therapy and participating institution. Therapy must begin within 6 weeks of surgery. Patients in the first group receive doxorubicin (or epirubicin) and cyclophosphamide every 28 days for a total of 4 cycles and oral tamoxifen daily for 5 years, beginning day 1 of chemotherapy. Patients in the second group receive the same chemotherapy with oral tamoxifen initiated on day 8 of the fourth chemotherapy cycle and continued for 5 years. Patients in the third group receive oral tamoxifen daily for 5 years. Patients in the fourth group are treated the same as the first group, only tamoxifen is replaced by toremifene. Patients in the fifth group are treated the same as the second group, only tamoxifen is replaced by toremifene. Patients in the sixth group receive oral toremifene daily for 5 years. The timing of optional radiotherapy for patients with less than total mastectomy in each group is based on institutional policy; radiotherapy is administered for 5-6 weeks to the remaining breast tissue, chest wall, and lung. Patients are followed every 3 months for 1 year, every 6 months for 2 years, and yearly thereafter.

PROJECTED ACCRUAL: 1,140 patients will be accrued over approximately 9 years, with 1 additional year of follow-up.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven stage T1-3, pN1, M0 carcinoma of the breast considered suitable for adjuvant treatment with endocrine therapy alone Estrogen receptor at least 10 fmol/mg cytosol protein or positive on immunohistochemical assay Potentially curative resection within 6 weeks of entry by one of the following: Total mastectomy with negative margins Breast-conserving procedure (lumpectomy or quadrantectomy) for tumors less than 5 cm Adequate re-resection or mastectomy within 4 weeks of initial surgery required if margins are positive after initial surgery Axillary clearance (not sampling) required at surgery, with at least 1 node positive upon histopathologic examination of at least 8 nodes Suspicious manifestations of metastatic disease (e.g., hot spots on bone scan, skeletal pain of unknown cause) must be proven benign No bilateral breast cancer Any mass in contralateral breast must be proven benign by biopsy

PATIENT CHARACTERISTICS: Age: 70 and under Sex: Women only Menopausal status: Peri/postmenopausal, i.e.: More than 6 months since last normal menstrual period (LNMP) with no prior hysterectomy and no hormone replacement therapy (HRT) Prior hysterectomy and no HRT and either age greater than 55 or age 55 or less with postmenopausal LH, FSH, and E2 levels On HRT and either age 50 or greater or LNMP more than 6 months prior to starting HRT Performance status: Not specified Hematopoietic: WBC greater than 4,000 Platelets greater than 100,000 Hepatic: Bilirubin less than 1.1 mg/dL (20 micromoles/L) AST less than 60 IU/L Renal: Creatinine less than 1.3 mg/dL (120 micromoles/L) Other: No nonmalignant systemic disease that would preclude protocol therapy or prolonged follow-up No psychiatric or addictive disorder that would preclude informed consent No prior or concurrent second malignancy except: Nonmelanomatous skin cancer Adequately treated in situ carcinoma of the cervix Geographically accessible for follow-up

PRIOR CONCURRENT THERAPY: No prior therapy for breast cancer other than potentially curative surgery (see Disease Characteristics)

Max Age: 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 452 (Actual)
Dates: Start 1993-05; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Overall survival | 17 years after randomization
  Time from randomization to death.

SECONDARY OUTCOMES:
Disease-free and systemic disease-free survival. | 17 years from randomization
  Time from randomization to recurrence, metastasis, appearance of a second primary tumor or death.
Quality of life | 17 years from randomization
  Quality of life will be assessed using QL Questionnaires of IBCSG.
Toxicity | 17 years after randomization
  Assessment of toxicity according to standard criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Edda Simoncini, MD, Study Chair — Spedali Civili di Brescia
Locations (20):
- Australia (5):
  - Newcastle Mater Misericordiae Hospital, Newcastle, New South Wales
  - Royal Prince Alfred Hospital, Sydney, Sydney, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Anti-Cancer Council of Victoria, Melbourne, Carlton South, Victoria
  - Sir Charles Gairdner Hospital, Perth, Perth, Western Australia
- Italy (5):
  - Centro di Riferimento Oncologico - Aviano, Aviano
  - Universita di Brescia, Brescia
  - Istituto Europeo Di Oncologia, Milan
  - Ospedale Civile Rimini, Rimini
  - Ospedale San Eugenio, Rome
- Auckland Adventist Hospital, Auckland, New Zealand
- Institute of Oncology, Ljubljana, Ljubljana, Slovenia
- Groote Schuur Hospital, Cape Town, Cape Town, South Africa
- Sahlgrenska University Hospital, Gothenburg (Goteborg), Sweden
- Switzerland (6):
  - University Hospital, Basel
  - Inselspital, Bern, Bern
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Hopital des Cadolles, Neuchatel, Neuchâtel
  - Kantonsspital - Saint Gallen, Sankt Gallen
  - Universitaetsspital, Zurich

REFERENCES:
- [Background] Gianni L, Gelber S, Ravaioli A, Price KN, Panzini I, Fantini M, Castiglione-Gertsch M, Pagani O, Simoncini E, Gelber RD, Coates AS, Goldhirsch A. Second non-breast primary cancer following adjuvant therapy for early breast cancer: a report from the International Breast Cancer Study Group. Eur J Cancer. 2009 Mar;45(4):561-71. doi: 10.1016/j.ejca.2008.10.011. Epub 2008 Dec 4. PMID 19062268
- [Background] Kenne Sarenmalm E, Oden A, Ohlen J, Gaston-Johansson F, Holmberg SB. Changes in health-related quality of life may predict recurrent breast cancer. Eur J Oncol Nurs. 2009 Dec;13(5):323-9. doi: 10.1016/j.ejon.2009.05.002. Epub 2009 Jul 12. PMID 19596212
- [Background] Pagani O, Gelber S, Simoncini E, Castiglione-Gertsch M, Price KN, Gelber RD, Holmberg SB, Crivellari D, Collins J, Lindtner J, Thurlimann B, Fey MF, Murray E, Forbes JF, Coates AS, Goldhirsch A; International Breast Cancer Study Group. Is adjuvant chemotherapy of benefit for postmenopausal women who receive endocrine treatment for highly endocrine-responsive, node-positive breast cancer? International Breast Cancer Study Group Trials VII and 12-93. Breast Cancer Res Treat. 2009 Aug;116(3):491-500. doi: 10.1007/s10549-008-0225-9. Epub 2008 Oct 25. PMID 18953651
- [Background] Pestalozzi BC, Zahrieh D, Mallon E, Gusterson BA, Price KN, Gelber RD, Holmberg SB, Lindtner J, Snyder R, Thurlimann B, Murray E, Viale G, Castiglione-Gertsch M, Coates AS, Goldhirsch A; International Breast Cancer Study Group. Distinct clinical and prognostic features of infiltrating lobular carcinoma of the breast: combined results of 15 International Breast Cancer Study Group clinical trials. J Clin Oncol. 2008 Jun 20;26(18):3006-14. doi: 10.1200/JCO.2007.14.9336. Epub 2008 May 5. PMID 18458044
- [Background] Keshaviah A, Dellapasqua S, Rotmensz N, Lindtner J, Crivellari D, Collins J, Colleoni M, Thurlimann B, Mendiola C, Aebi S, Price KN, Pagani O, Simoncini E, Castiglione Gertsch M, Gelber RD, Coates AS, Goldhirsch A. CA15-3 and alkaline phosphatase as predictors for breast cancer recurrence: a combined analysis of seven International Breast Cancer Study Group trials. Ann Oncol. 2007 Apr;18(4):701-8. doi: 10.1093/annonc/mdl492. Epub 2007 Jan 20. PMID 17237474
- [Background] Gianni L, Panzini I, Li S, Gelber RD, Collins J, Holmberg SB, Crivellari D, Castiglione-Gertsch M, Goldhirsch A, Coates AS, Ravaioli A; International Breast Cancer Study Group (IBCSG). Ocular toxicity during adjuvant chemoendocrine therapy for early breast cancer: results from International Breast Cancer Study Group trials. Cancer. 2006 Feb 1;106(3):505-13. doi: 10.1002/cncr.21651. PMID 16369994
- [Background] International Breast Cancer Study Group; Pagani O, Gelber S, Price K, Zahrieh D, Gelber R, Simoncini E, Castiglione-Gertsch M, Coates AS, Goldhirsch A. Toremifene and tamoxifen are equally effective for early-stage breast cancer: first results of International Breast Cancer Study Group Trials 12-93 and 14-93. Ann Oncol. 2004 Dec;15(12):1749-59. doi: 10.1093/annonc/mdh463. PMID 15550579